CLINICAL TRIAL: NCT02005198
Title: Assessing the Minimal Important Difference (MID) of the Treatment Related Impact Measure-Adult Growth Hormone Deficiency (TRIM-AGHD)
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN8640-4123; U1111-1146-1750 (Other: WHO)
Record Dates: First submitted 2013-12-03; First posted 2013-12-09 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Growth Hormone Disorder; Adult Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Survey
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — Subject will only fill out a questionnaire when entering the non-interventional study

SUMMARY:
This study is conducted in the United States of America (USA). The aim of the study is to assess the minimal important difference (MID) of the TRIM-AGHD.

ELIGIBILITY:
Inclusion Criteria:

* Able to speak read and write English
* GHD (Growth Hormone Deficiency) treatment naïve which is defined as not being on a prescription treatment for their GHD currently and for at least 6 months
* Beginning a new prescription GHD treatment and expected to be on this treatment for GHD for a minimum of 6 months
* GHD of either one of the following criteria: a) Adult onset: subjects who have GHD, either alone or associated with multiple hormone deficiencies (hypopituitarism), as a result of pituitary disease, hypothalamic disease, surgery, radiation therapy, or traumatic brain injury (TBI), b) Childhood Onset: Subjects who were growth hormone deficient during childhood as a result of congenital, genetic, acquired, or idiopathic causes
* Confirmed diagnosis of growth hormone deficiency (if a subject satisfies any one of the three following criteria): a) For the insulin tolerance test (ITT) or glucagon test both performed within the last five years: the validated cut-off for GHD in adults is a peak GH response of below 3.0 ng/mL (3 microg/L), b) For growth hormone releasing hormone (GHRH) +Arginine test performed within the last five years: for those subjects with a body mass index (BMI) below 25 kg/m^2, a peak GH below 11 ng/mL (microg /L); for BMI 25-30 kg/m^2, a peak GH below 8 ng/mL (8 microg/L); for BMI above 30 kg/m^2, a peak GH below 4 ng/mL 341 (4 microg/L ), c) Three or more pituitary hormone deficiencies at screening
* Informed consent obtained before any study-related activities. (Study-related activities are any procedure related to recording of data according to the protocol)

Exclusion Criteria:

* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
* Patients who have been on a prescription medication for treatment of GHD in past 6 months
* Patients with a total Beck Depression Inventory II (BDI-II) score greater than 25
* Females who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods (adequate contraceptive measures as required by local law or practice)
* Acute severe illness associated with weight loss in the last 6 months (defined as a loss of more than 5.0% total body weight)
* Active Cushings syndrome within the last 24 months
* Subject with overt diabetes mellitus
* Previous participation in this study

Ages: 23 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a diagnosis of growth hormone deficiency (GHD), naïve to treatment currently and for at least 6 months prior, who are beginning a new prescription treatment for their GHD. Patients will be selected by sites as per inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2014-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Changes in CGI (Clinician Global Impression Scale) | After the physician scheduled visits closest to week 8 and week 26 after initiation of treatment
Changes in PGI (Patient Global Impression Scale) | After the physician scheduled visits closest to week 8 and week 26 after initiation of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Princeton, New Jersey, United States

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com